CLINICAL TRIAL: NCT06308406
Title: A Phase Ib/II Clinical Study of HRS-1167 in Combination With Bevacizumab in Patients With Recurrent Ovarian Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-1167-201-Bev
Record Dates: First submitted 2024-02-26; First posted 2024-03-13 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-02

CONDITIONS: Recurrent Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-1167 in combination with bevacizumab in patients with recurrent ovarian cancer (Experimental)
  Interventions: Drug: Bevacizumab； HRS-1167

INTERVENTIONS:
Drug: Bevacizumab； HRS-1167 — Bevacizumab: injection, 100mg(4mL), intravenous infusion HRS-1167: Tablets, 25mg/tablet, oral

SUMMARY:
This study is a multicenter, open-label Phase Ib/II clinical trial to observe and evaluate the safety, tolerability and pharmacokinetics of HRS-1167 in combination with bevacizumab in patients with recurrent ovarian cancer mechanical characterization and preliminary evaluation of the efficacy of HRS-1167 in combination with bevacizumab in patients with recurrent ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily join this study, sign the informed consent form, have good compliance, and be able to cooperate with the follow-up.
2. Age 18~75 years old.
3. Cytologically or histologically confirmed diagnosis of recurrent epithelial ovarian, fallopian tube, or primary peritoneum cancer.
4. Patient has been previously treated with a platinum-containing regimen and has been treated with a platinum-based regimen during the last dose of platinum-based therapy (self-treatment initiation to within 1 month after the last dose) efficacy is non-PD, 6 months after the end of treatment (183 disease progression or recurrence within calendar days, and the number of lines of systemic therapy after platinum resistance ≤1 line.
5. At least one measurable lesion per RECIST v1.1 criteria.
6. ECOG PS score: 0-1 points.
7. Expected survival period ≥ 3 weeks.
8. Good level of organ function.
9. Subjects of childbearing potential who need to use highly effective contraception from the time of signing informed to 210 days after the last dose of trial drug; Subjects of childbearing potential must have a negative serum HCG within 7 days prior to the first dose and must be non-lactating.

Exclusion Criteria:

1. Those who have received chemotherapy, immune checkpoint inhibitors, major surgical operations, anti-tumor vaccines within 4 weeks before the first dose; Those who have received palliative radiotherapy within 2 weeks prior to the first dose; Oral molecularly targeted therapy (including other clinical trial targeted agents) 5 drug half-lives or 4 weeks (whichever is shorter) < from the first study dose; Those who have received a live vaccine within 4 weeks prior to the first dose or possibly during the study.
2. Toxicity due to prior antineoplastic therapy has not recovered according to NCI-CTCAE v5.0 grade≤ Level 1.
3. Subject has previous or concurrent other malignancies.
4. Subject has carcinomatous meningitis, or has untreated central nervous system metastases.
5. Imaging shows tumor invasion of large blood vessels or unclear demarcation from blood vessels; or the investigator judges that the patient's tumor has a high possibility of invading important blood vessels and causing fatal hemorrhage during treatment.
6. Cancerous ascites and pleural effusion with clinical symptoms, requiring puncture and drainage; or those who have received ascites, pleural effusion drainage within 14 days before the first dose of the drug.
7. Severe bone injury due to tumor bone metastases, including severe bone pain with poor control, pathological fractures of important sites and spinal cord that have occurred within the last 6 months or are expected to occur in the near future oppression, etc.
8. Previous or current interstitial pneumonitis/interstitial lung disease (except for those with radiographic changes only), pneumonia requiring systemic treatment with glucocorticoids (such as radiation pneumonitis, etc.); Current active pneumonitis or those with severe impairment of lung function confirmed by pulmonary function tests.
9. People who are known to be allergic to bevacizumab or have had a severe allergic reaction to other monoclonal antibodies.
10. Those with active tuberculosis; Those who have been adequately treated before the first dose and have discontinued anti-tuberculosis therapy for ≥ 3 months can be enrolled.
11. Have hypertension that is not well controlled with antihypertensive medication (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 90 mmHg); Previous hypertensive crisis or hypertensive sex encephalopathy.
12. Have clinical symptoms or disease of the heart that are not well controlled.
13. Coagulation abnormalities, bleeding tendency, or those receiving thrombolytic or anticoagulant therapy are allowed to receive low-dose low-molecular-weight heparin or oral aspirin prophylactic anticoagulation therapy during the trial.
14. NCI-CTCAE v5.0 grade ≥2 bleeding events within 4 weeks prior to the first dose, including but not limited to hemoptysis (hemoptysis in a single episode ≥2mL), vaginal bleeding, gastrointestinal bleeding, etc.
15. Experienced arterior/venous thrombotic event within 6 months prior to the first dose.
16. Patients with gastrointestinal perforation or fistula (except artificial fistula), urethral fistula, intra-abdominal abscess, intestinal obstruction, or those requiring parenteral nutrition within 3 months prior to the first dose.
17. Those who are unable to swallow tablets normally, or have abnormal gastrointestinal function, which may affect drug absorption as judged by the investigator.
18. Subjects who have had a serious infection within 1 month before the first dose, including but not limited to infectious complications requiring hospitalization, bacteremia, severe pneumonia, etc.; Subjects with any active infection requiring intravenous system therapy, or who have a progeny during the screening period, prior to the first dose 38.5°C due to unknown fever>; Those who have used antibiotics within 2 weeks before the first dose.
19. Known history of positive human immunodeficiency virus (HIV) test; Known active hepatitis.
20. Treatment with a strong inhibitor of CYP3A4, CYP2D6, P-gp, or BCRP, <5 drug half-lives or 14 days from the date of first dose; Treatment with the above enzyme strong inducers was 28 days < the first dose.
21. As judged by the investigator, there are other factors that may affect the results of the study or cause the study to be terminated halfway, such as alcoholism, drug abuse, other serious diseases (such as severe diabetes, thyroid disease, spinal cord compression, superior vena cava syndrome, psychiatric diseases) that require concomitant treatment, serious laboratory test abnormalities, accompanied by family or social factors, which will affect the safety of the subjects.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The number of subjects with dose-limiting toxicity (DLT) | From first dose of study treatment until the end of Cycle 1（up to 21 days）
Determination of Recommended Phase II dose (RP2D) | From first dose of study treatment until the end of Cycle 1（up to 21 days）

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From time of first dose of HRS-1167 or Bevacizumab until the date of objective disease progression or death (up to 24 months)]
  The percentage of participants with a confirmed CR or PR according to RECIST v1.1 criteria.
Disease Control Rate (DCR) | From time of first dose of HRS-1167 or Bevacizumab until the date of objective disease progression or death (up to 24 months)
  The percentage of participants who have a best objective response of confirmed CR or PR or who have SD for at least 15 weeks after start of treatment
Duration of Response (DoR) | From time of first dose of HRS-1167 or Bevacizumab until the date of objective disease progression or death (up to 24 months)
  The time from the date of first response until date of disease progression or death in the absence of disease progression.
Progression free Survival (PFS) | From time of fist dose of HRS-1167 or Bevacizumab until the date of objective disease progression or death (up to 24 months)
  Progression-free survival is defined as the time from the start of treatment until the date of objective disease progression or death
Overall Survival (OS) | From time of first dose of HRS-1167 or Bevacizumab until the date of death (up to 24 months)
  The time until death due to any cause.
Time To Response(TTR) | From time of first dose of HRS-1167 or Bevacizumab until the date of objective disease progression or death (up to 24 months)
  Time from C1D1 to complete or partial response, according to RECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong First Medical University Affiliated Cancer Hospital, Jinan, Shangdong
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided